CLINICAL TRIAL: NCT04724980
Title: A Phase 1/2 Study of Adjuvant PRGN-2012 in Adult Patients With Recurrent Respiratory Papillomatosis
Brief Title: Adjuvant PRGN-2012 in Adult Patients With Recurrent Respiratory Papillomatosis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Precigen, Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210013; 21-C-0013
Record Dates: First submitted 2021-01-23; First posted 2021-01-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Respiratory Papillomatosis; Papillomavirus Infections; Papillomaviridae
Keywords: Human Papilloma Virus; Dose escalation; laryngotracheal disease; papillomatous disease
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Arm1: Dose level 1: 1x10^11 (Phase I) Arm2: Dose level 2: 5x10^11 (Phase I) Amr3: Dose level 3: 5x10^11 (Phase II)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I; Dose Level 1 (Experimental): A standard dose escalation design was used to evaluate PRGN-2012 at a dose level of 1 × 10^11
  Interventions: Drug: PRGN-2012 - Phase I; Dose Level 1
- Phase I; Dose Level 2 (Experimental): A standard dose escalation design was used to evaluate PRGN-2012 at a dose level of 5 × 10^11
  Interventions: Drug: PRGN-2012 - Phase I; Dose Level 2
- Phase II; Dose Level 2 (Experimental): A dose of 5 x 10^11 PU was established as the RP2D, and the Phase 2 portion was implemented. The Phase 2 portion is designed as a dose expansion study, where patients were treated at the RP2D to evaluate the safety and efficacy of PRGN-2012.
  Interventions: Drug: PRGN-2012 - Phase II; Dose Level 2

INTERVENTIONS:
Drug: PRGN-2012 - Phase I; Dose Level 1 — In Phase 1, dose level 1 of the clinical trial, PRGN-2012 is administered at 1 × 10^11 particle units as adjuvant therapy prior to standard debulking surgery.
  Arms: Phase I; Dose Level 1
Drug: PRGN-2012 - Phase I; Dose Level 2 — In Phase 1, dose level 2 of the clinical trial, PRGN-2012 is administered at 5 × 10^11 particle units as adjuvant therapy prior to standard debulking surgery.
  Arms: Phase I; Dose Level 2
Drug: PRGN-2012 - Phase II; Dose Level 2 — The Phase 2 portion is designed as a dose expansion study where patients are treated at the RP2D of 5 x 10^11 PU.
  Arms: Phase II; Dose Level 2

SUMMARY:
This is a Phase 1/2 study in patients with a Recurrent Respiratory Papillomatosis (RRP) disease burden that requires repeated surgical procedures for management. RRP is a rare disease caused by the human papillomavirus (HPV). Participants with a pathologically confirmed diagnosis of papilloma and a clinical diagnosis of RRP will be screened for this protocol.

DETAILED DESCRIPTION:
This is a nonrandomized, Phase 1/2 safety and tolerability study. The safety and tolerability of PRGN-2012 will be assessed following two different dose levels during the Phase 1 dose escalation trial. In the Phase 2 portion of the study, treatment with PRGN-2012 at the recommended Phase 2 dose (RP2D) will be used to determine safety and efficacy of PRGN-2012.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18 years and older
* Clinical diagnosis of RRP

  * Histological diagnosis of papilloma confirmed by pathology report from a CLIA-certified (or comparable) laboratory
  * Presence of laryngotracheal papillomas with or without pulmonary RRP
  * A history of 3 or more interventions in the last 12 months for control of RRP
  * Clinical performance status of ECOG of 0-1
* Willing to undergo endoscopic evaluation and operative interventions with biopsies in compliance with this protocol
* No systemic therapy for RRP for at least 3 half-lives of the prior drug(s). A 30-day washout is required for systemic bevacizumab treatment
* Participants who have received prior immunotherapy for RRP are permitted
* Participants must have adequate organ and marrow function as defined below:
* Sexually active subjects (men and women) of reproductive potential must agree to use two methods of contraception: one highly effective and one other effective method throughout vaccine treatment and for at least 120 days after vaccine treatment. Highly effective methods are defined as: Intrauterine device (IUD), hormonal (birth control pills, injections, implants), tubal ligation, and partner's vasectomy; other effective methods are defined as a latex condom, diaphragm, and cervical cap.
* Seronegative for hepatitis B antigen, positive hepatitis B tests can be further evaluated by confirmatory tests (Hep B DNA quant, HBV viral load), and if confirmatory tests are negative, the participant can be enrolled.
* Seronegative for hepatitis C antibody unless antigen negative. If the hepatitis C antibody test is positive, then participants must be tested for the presence of antigen by Hep C RNA quant, HCV viral load, and be HCV RNA negative
* All participants must have the ability to understand and willingness to sign a written informed consent

EXCLUSION CRITERIA:

* A history of surgical debridement of papillomas such that in the opinion of the study team a participant is unlikely to be able to safely have a six-week interval between clinically indicated interventions.
* History of significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (greater than or equal to New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Any severe acute or chronic medical or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior, liver disease, lung disease (with the exception of what is specified in the inclusion criteria) , or laboratory abnormalities that, in the opinion of the investigators, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results and in the judgment of the investigator, would make the participant inappropriate for entry into this study. Participants with mild to moderate asthma or chronic obstructive pulmonary disease (COPD) well controlled with oral or inhaled medications are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled, topical intranasal or intro-ocular steroids, and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Participants who are receiving any other investigational agents
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 5.0; however, alopecia, sensory neuropathy Grade less than or equal to 2 or other Grade less than or equal to 2 AEs not constituting a safety risk based on investigator's judgment are acceptable.
* Known alcohol or drug abuse.
* Participant, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* History of allergy to study drug components.
* Pregnant women are excluded from this study because PRGN-2012 is an agent with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PRGN-2012, breastfeeding should be discontinued if the mother is treated with PRGN-2012. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Determine the percentage of subjects with a complete response following treatment with PRGN-2012 | 1 year
  A complete response is defined as no requirement for surgical intervention in the 12 months after treatment
Determine the incidence of dose limiting toxicities to evaluate safety and identify RP2D of PRGN-2012 | 28 days
  The incidence of dose limiting toxicities in Phase 1 will be reported per dose level. The dose level at which less than or equal to 1 out of 6 patients experience DLT will be identified as a RP2D.

SECONDARY OUTCOMES:
Safety of PRGN 2012 at RP2D | 1 year
  Systemic toxicity will be assessed through the capture of Treatment Emergent Adverse Events ( TEAEs) at Phase 1 and Phase 2 patients. The severity of the TEAEs will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 scale.
Immune Responses | 1 year
  Change in HPV-specific T cells post-treatment compared to baseline
Change in RRP Staging Assessment Scores Over Time | 1 year
  Absolute and percentage change from baseline in Derkay score over time following initiation of PRGN-2012 treatment
Change in Vocal Function Scores over Time | 1 year
  Absolute and percentage change from baseline in VHI-10 score over time following initiation of PRGN-2012 treatment
Time to recurrence of papillomatous disease after completion of treatment | 1 year
  Time to recurrence of papillomatous disease after completion of treatment will be recorded. Time from completion of treatment to first surgery will be assessed.
Percentage of subjects with reduction in number of surgeries after completion of treatment | 1 year
  The number of surgeries in the 12 months post-treatment will be compared to the number of surgeries in the 12 months pre-treatment to identify subjects that have a reduction in the number of surgeries.
Number of surgery during the 12 months pre and 12 months post treatment | 1 year
  The number of surgeries in the 12 months post-treatment will be compared to the number of surgeries in the 12 months pre-treatment.
Overall Response Rate | 1 year
  Determine the percentage of subjects with at least a 50% decrease in the number of surgeries during the 12 month period following completion of PRGN-2012 treatment as compared to the number of surgeries during the 12 months prior to PRGN-2012 treatment initiation.
Rate of pulmonary RRP partial response in participants with pulmonary disease | 1 year
  The fraction of participants with a pulmonary RRP partial response will be reported in all treated pulmonary participants.
Rate of pulmonary RRP complete response in participants with pulmonary disease | 1 year
  The fraction of participants with a pulmonary RRP complete response will be reported in all treated pulmonary participants.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lankford, PhD, Study Director — Precigen, Inc
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Norberg SM, Valdez J, Napier S, Kenyon M, Ferraro E, Wheatley M, Parsons-Wandell L, Doran SL, Lankford A, Sabzevari H, Brough DE, Schlom J, Gulley JL, Allen CT. PRGN-2012 gene therapy in adults with recurrent respiratory papillomatosis: a pivotal phase 1/2 clinical trial. Lancet Respir Med. 2025 Apr;13(4):318-326. doi: 10.1016/S2213-2600(24)00368-0. Epub 2025 Jan 21. PMID 39855244
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0013.html